CLINICAL TRIAL: NCT01154218
Title: A Phase 1, Single Dose Bioequivalence And Food Effect Study In Healthy Volunteers Comparing The Commercial Image Capsules To The Immediate Release Tablets And Powder In Capsule Formulations Of Crizotinib (PF-02341066), And The Commercial Image Capsule In The Fasted To Fed State
Brief Title: Bioequivalence And Food Effect Study Comparing The Commercial Formulation Of Crizotinib To Its Clinical Study Formulations And Commercial Formulation With Or Without Food In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: A8081011
Record Dates: First submitted 2010-06-29; First posted 2010-06-30 (Estimated); Results first posted 2011-10-19 (Estimated); Last update posted 2011-10-24 (Estimated); Status verified 2011-10

CONDITIONS: Healthy
Keywords: bioequivalence; food effect; pharmacokinetics; crizotinib
MeSH Terms: interventions — Crizotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): All subjects will receive four treatments in one of the indicated orders:
  A-B-C-D, B-D-A-C, C-A-D-B, D-C-B-A
  Interventions: Drug: crizotinib

INTERVENTIONS:
Drug: crizotinib — Treatment A (Reference 1): a 250 mg single dose of crizotinib administered in a fasted state as 1 × 50-mg IRT and 2 × 100-mg IRTs.
  Treatment B (Reference 2): a 250 mg single dose of crizotinib administered in a fasted state as 1 × 50-mg PIC and 2 × 100 mg PICs.
  Treatment C (Test for BE, Reference for Food Effect): a 250 mg single dose of crizotinib administered in a fasted state as 1 × 250-mg CIC.
  Treatment D (Test High Fat): a 250 mg single dose of crizotinib administered with a high-fat meal as 1 × 250-mg CIC

SUMMARY:
The purpose of this study is to demonstrate bioequivalence of the Commercial Image Capsule (CIC) relative to the Immediate Release Tablet (IRT) of crizotinib, bioequivalence of CIC relative to Powder in Capsule (PIC) of crizotinib, and lack of an effect of high fat meal on the pharmacokinetics (PK) of crizotinib when administered as CIC Formulation in healthy volunteers.

DETAILED DESCRIPTION:
The purpose of this study is to demonstrate bioequivalence of the CIC relative to IRT and CIC relative to PIC, and lack of an effect of food on the PK of crizotinib in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female of non-childbearing potential subjects between the ages of 18 and 55 years, inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests).
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m^2; and a total body weight >50 kg (110 lbs)

Exclusion Criteria:

* Subjects who are smoking, or with evidence of disease, conditions affecting absorption, treatment with other investigational drug within 30 days, history of regular alcohol consumption, use of prescription, nonprescription drugs and dietary supplement within 7 days, or blood donation of 500 mL within 56 days.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2010-08; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8081011&StudyName=Bioequivalence%20And%20Food%20Effect%20Study%20Comparing%20The%20Commercial%20Formulation%20Of%20Crizotinib%20To%20Its%20Clinical%20Study%20Formulations%20And%20Commercial%20

RESULTS

PARTICIPANT FLOW:
Groups:
- Crizotinib 250 mg IRT Fasted, PIC Fasted, CIC Fasted, CIC Fed: Single oral dose of crizotinib 250 milligram (mg) immediate release tablet (IRT) in fasted state in first intervention period; followed by single oral dose of crizotinib 250 mg powder in capsule (PIC) in fasted state in second intervention period; followed by single oral dose of crizotinib 250 mg commercial image capsule (CIC) in fasted state in third intervention period; and single oral dose of crizotinib 250 mg CIC in fed state in fourth intervention period. A washout period of at least 14 days was maintained between each period.
- Crizotinib 250 mg PIC Fasted, CIC Fed, IRT Fasted, CIC Fasted: Single oral dose of crizotinib 250 mg PIC in fasted state in first intervention period; followed by single oral dose of crizotinib 250 mg CIC in fed state in second intervention period; followed by single oral dose of crizotinib 250 mg IRT in fasted state in third intervention period; and single oral dose of crizotinib 250 mg CIC in fasted state in fourth intervention period. A washout period of at least 14 days was maintained between each period.
- Crizotinib 250 mg CIC Fasted, IRT Fasted, CIC Fed, PIC Fasted: Single oral dose of crizotinib 250 mg CIC in fasted state in first intervention period; followed by single oral dose of crizotinib 250 mg IRT in fasted state in second intervention period; followed by single oral dose of crizotinib 250 mg CIC in fed state in third intervention period; and single oral dose of crizotinib 250 mg PIC in fasted state in fourth intervention period. A washout period of at least 14 days was maintained between each period.
- Crizotinib 250 mg CIC Fed, CIC Fasted, PIC Fasted, IRT Fasted: Single oral dose of crizotinib 250 mg CIC in fed state in first intervention period; followed by single oral dose of crizotinib 250 mg CIC in fasted state in second intervention period; followed by single oral dose of crizotinib 250 mg PIC in fasted state in third intervention period; and single oral dose of crizotinib 250 mg IRT in fasted state in fourth intervention period. A washout period of at least 14 days was maintained between each period.
Period: First Intervention Period
Arm/Group | Crizotinib 250 mg IRT Fasted, PIC Fasted, CIC Fasted, CIC Fed | Crizotinib 250 mg PIC Fasted, CIC Fed, IRT Fasted, CIC Fasted | Crizotinib 250 mg CIC Fasted, IRT Fasted, CIC Fed, PIC Fasted | Crizotinib 250 mg CIC Fed, CIC Fasted, PIC Fasted, IRT Fasted
Started | 9 | 9 | 9 | 9
Completed | 9 | 9 | 9 | 9
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period (at Least 14 Days)
Arm/Group | Crizotinib 250 mg IRT Fasted, PIC Fasted, CIC Fasted, CIC Fed | Crizotinib 250 mg PIC Fasted, CIC Fed, IRT Fasted, CIC Fasted | Crizotinib 250 mg CIC Fasted, IRT Fasted, CIC Fed, PIC Fasted | Crizotinib 250 mg CIC Fed, CIC Fasted, PIC Fasted, IRT Fasted
Started | 9 | 9 | 9 | 9
Completed | 9 | 9 | 9 | 9
Not Completed | 0 | 0 | 0 | 0
Period: Second Intervention Period
Arm/Group | Crizotinib 250 mg IRT Fasted, PIC Fasted, CIC Fasted, CIC Fed | Crizotinib 250 mg PIC Fasted, CIC Fed, IRT Fasted, CIC Fasted | Crizotinib 250 mg CIC Fasted, IRT Fasted, CIC Fed, PIC Fasted | Crizotinib 250 mg CIC Fed, CIC Fasted, PIC Fasted, IRT Fasted
Started | 9 | 9 | 9 | 9
Completed | 9 | 9 | 9 | 9
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period (at Least 14 Days)
Arm/Group | Crizotinib 250 mg IRT Fasted, PIC Fasted, CIC Fasted, CIC Fed | Crizotinib 250 mg PIC Fasted, CIC Fed, IRT Fasted, CIC Fasted | Crizotinib 250 mg CIC Fasted, IRT Fasted, CIC Fed, PIC Fasted | Crizotinib 250 mg CIC Fed, CIC Fasted, PIC Fasted, IRT Fasted
Started | 9 | 9 | 9 | 9
Completed | 9 | 9 | 9 | 9
Not Completed | 0 | 0 | 0 | 0
Period: Third Intervention Period
Arm/Group | Crizotinib 250 mg IRT Fasted, PIC Fasted, CIC Fasted, CIC Fed | Crizotinib 250 mg PIC Fasted, CIC Fed, IRT Fasted, CIC Fasted | Crizotinib 250 mg CIC Fasted, IRT Fasted, CIC Fed, PIC Fasted | Crizotinib 250 mg CIC Fed, CIC Fasted, PIC Fasted, IRT Fasted
Started | 9 | 9 | 9 | 9
Completed | 9 | 8 | 9 | 9
Not Completed | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0
Period: Washout Period (at Least 14 Days)
Arm/Group | Crizotinib 250 mg IRT Fasted, PIC Fasted, CIC Fasted, CIC Fed | Crizotinib 250 mg PIC Fasted, CIC Fed, IRT Fasted, CIC Fasted | Crizotinib 250 mg CIC Fasted, IRT Fasted, CIC Fed, PIC Fasted | Crizotinib 250 mg CIC Fed, CIC Fasted, PIC Fasted, IRT Fasted
Started | 9 | 8 | 9 | 9
Completed | 9 | 8 | 9 | 8
Not Completed | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Period: Fourth Intervention Period
Arm/Group | Crizotinib 250 mg IRT Fasted, PIC Fasted, CIC Fasted, CIC Fed | Crizotinib 250 mg PIC Fasted, CIC Fed, IRT Fasted, CIC Fasted | Crizotinib 250 mg CIC Fasted, IRT Fasted, CIC Fed, PIC Fasted | Crizotinib 250 mg CIC Fed, CIC Fasted, PIC Fasted, IRT Fasted
Started | 9 | 8 | 9 | 8
Completed | 8 | 8 | 9 | 8
Not Completed | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes participants randomized to receive any treatment (crizotinib 250 mg IRT fasted first, crizotinib 250 mg PIC fasted first, crizotinib 250 mg CIC fasted first and crizotinib 250 mg CIC fed).
Arm/Group | Entire Study Population
Number analyzed (Participants) | 36
Age Continuous [Mean (Standard Deviation); unit: years] | 38.9 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 36

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUC [0 - ∞])
Description: AUC (0-∞) = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-∞). It is obtained from AUC (0-t) plus AUC (t-∞).
Time Frame: 0 (pre-dose), 1, 2, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96 and 144 hours (hrs) post crizotinib dose
Population: Pharmacokinetic (PK) parameter analysis population included all randomized and treated participants who had at least 1 of the PK parameters of primary interest in at least 1 treatment period.
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Groups:
- Crizotinib IRT Fasted: Single oral dose of crizotinib 250 mg IRT (Treatment A [Reference 1]) in fasted state in any intervention period.
- Crizotinib PIC Fasted: Single oral dose of crizotinib 250 mg PIC (Treatment B [Reference 2]) in fasted state in any intervention period.
- Crizotinib CIC Fasted: Single oral dose of crizotinib 250 mg CIC (Treatment C [Test for bioequivalence (BE), Reference for Food effect]) in fasted state in any intervention period.
- Crizotinib CIC Fed: Single oral dose of crizotinib 250 mg CIC (Treatment D [Test High Fat]) in fed state in any intervention period.
Arm/Group | Crizotinib IRT Fasted | Crizotinib PIC Fasted | Crizotinib CIC Fasted | Crizotinib CIC Fed
Number analyzed (Participants) | 35 | 35 | 35 | 36
ng*hr/mL | 2890.0 (1021.8) | 2665.0 (1190.4) | 2887.0 (1109.6) | 2475.0 (1037.7)
Statistical Analysis 1: Comparison: Crizotinib IRT Fasted vs Crizotinib CIC Fasted; Natural log transformed AUC (0-∞) of crizotinib was analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. The adjusted mean differences and 90% confidence intervals (CIs) for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios; Test type: Superiority or Other; Ratio of Adjusted Means = 99.56, 90% CI 2-sided [91.49 to 108.33]
Statistical Analysis 2: Comparison: Crizotinib PIC Fasted vs Crizotinib CIC Fasted; Natural log transformed AUC (0-∞) of crizotinib was analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. The adjusted mean differences and 90% CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios; Test type: Superiority or Other; Ratio of Adjusted means = 106.93, 90% CI 2-sided [98.26 to 116.35]
Statistical Analysis 3: Comparison: Crizotinib CIC Fasted vs Crizotinib CIC Fed; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; Ratio of Adjusted Means = 85.76, 90% CI 2-sided [78.88 to 93.25]

2. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast)
Description: Area under the plasma concentration time-curve from zero (pre-dose) to the last measured concentration (AUClast).
Time Frame: 0 (pre-dose), 1, 2, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96 and 144 hrs post crizotinib dose
Population: PK parameter analysis population included all randomized and treated participants who had at least 1 of the PK parameters of primary interest in at least 1 treatment period.
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Crizotinib IRT Fasted | Crizotinib PIC Fasted | Crizotinib CIC Fasted | Crizotinib CIC Fed
Number analyzed (Participants) | 35 | 35 | 35 | 36
ng*hr/mL | 2763.0 (989.0) | 2531.0 (1158.0) | 2761.0 (1078.4) | 2359.0 (1013.0)
Statistical Analysis 1: Comparison: Crizotinib IRT Fasted vs Crizotinib CIC Fasted; Natural log transformed AUClast of crizotinib was analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. The adjusted mean differences and 90% CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios; Test type: Superiority or Other; Ratio of Adjusted means = 99.60, 90% CI 2-sided [91.30 to 108.66]
Statistical Analysis 2: Comparison: Crizotinib PIC Fasted vs Crizotinib CIC Fasted; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Ratio of Adjusted means = 107.56, 90% CI 2-sided [98.58 to 117.35]
Statistical Analysis 3: Comparison: Crizotinib CIC Fasted vs Crizotinib CIC Fed; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Ratio of Adjusted means = 85.52, 90% CI 2-sided [78.45 to 93.22]

3. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax)
Time Frame: 0 (pre-dose), 1, 2, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96 and 144 hrs post crizotinib dose
Population: as for outcome 2
Measure: Median (Full Range); unit: hr
Arm/Group | Crizotinib IRT Fasted | Crizotinib PIC Fasted | Crizotinib CIC Fasted | Crizotinib CIC Fed
Number analyzed (Participants) | 35 | 35 | 35 | 36
hr | 5.00 [1.00 to 8.00] | 5.00 [2.00 to 6.00] | 5.00 [2.00 to 6.00] | 5.00 [1.00 to 8.00]

4. Secondary Outcome: Plasma Decay Half Life (t1/2)
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: 0 (pre-dose), 1, 2, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96 and 144 hrs post crizotinib dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Crizotinib IRT Fasted | Crizotinib PIC Fasted | Crizotinib CIC Fasted | Crizotinib CIC Fed
Number analyzed (Participants) | 35 | 35 | 35 | 36
hr | 34.62 (4.13) | 35.28 (6.39) | 34.85 (4.94) | 35.41 (5.49)

5. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Time Frame: 0 (pre-dose), 1, 2, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96 and 144 hrs post crizotinib dose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Crizotinib IRT Fasted | Crizotinib PIC Fasted | Crizotinib CIC Fasted | Crizotinib CIC Fed
Number analyzed (Participants) | 35 | 35 | 35 | 36
ng/mL | 126.00 (36.58) | 119.30 (50.88) | 135.00 (47.84) | 116.10 (45.58)
Statistical Analysis 1: Comparison: Crizotinib IRT Fasted vs Crizotinib CIC Fasted; Natural log transformed Cmax of crizotinib was analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. The adjusted mean differences and 90% CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios; Test type: Superiority or Other; Ratio of Adjusted Means = 106.97, 90% CI 2-sided [96.55 to 118.51]
Statistical Analysis 2: Comparison: Crizotinib PIC Fasted vs Crizotinib CIC Fasted; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; Ratio of Adjusted Means = 111.32, 90% CI 2-sided [100.47 to 123.33]
Statistical Analysis 3: Comparison: Crizotinib CIC Fasted vs Crizotinib CIC Fed; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; Ratio of Adjusted Means = 86.22, 90% CI 2-sided [77.89 to 95.43]

6. Secondary Outcome: Apparent Oral Clearance (CL/F)
Description: Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the body. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed.
Time Frame: 0 (pre-dose), 1, 2, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96 and 144 hrs post crizotinib dose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: L/hr
Arm/Group | Crizotinib IRT Fasted | Crizotinib PIC Fasted | Crizotinib CIC Fasted | Crizotinib CIC Fed
Number analyzed (Participants) | 35 | 35 | 35 | 36
L/hr | 86.49 (30.42) | 93.78 (49.80) | 86.57 (53.63) | 101.00 (38.60)

7. Secondary Outcome: Apparent Volume of Distribution (Vz/F)
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Time Frame: 0 (pre-dose), 1, 2, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96 and 144 hrs post crizotinib dose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: L
Arm/Group | Crizotinib IRT Fasted | Crizotinib PIC Fasted | Crizotinib CIC Fasted | Crizotinib CIC Fed
Number analyzed (Participants) | 35 | 35 | 35 | 36
L | 4290.0 (1672.4) | 4703.0 (2874.7) | 4313.0 (3880.9) | 5096.0 (2302.0)

8. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) for Crizotinib Metabolite (PF-06260182)
Description: Area under the plasma concentration time-curve from zero (pre-dose) to the last measured concentration (AUClast) of Crizotinib metabolite (PF-06260182).
Time Frame: 0 (pre-dose), 1, 2, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96 and 144 hrs post crizotinib dose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Crizotinib IRT Fasted | Crizotinib PIC Fasted | Crizotinib CIC Fasted | Crizotinib CIC Fed
Number analyzed (Participants) | 35 | 35 | 35 | 36
ng*hr/mL | 432.20 (219.76) | 391.20 (255.12) | 436.90 (246.34) | 325.00 (192.81)
Statistical Analysis 1: Comparison: Crizotinib IRT Fasted vs Crizotinib CIC Fasted; Natural log transformed AUClast of PF-06260182 was analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. The adjusted mean differences and 90% CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios; Test type: Superiority or Other; Ratio of Adjusted means = 100.03, 90% CI 2-sided [90.16 to 110.97]
Statistical Analysis 2: Comparison: Crizotinib PIC Fasted vs Crizotinib CIC Fasted; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; Ratio of Adjusted means = 108.85, 90% CI 2-sided [98.11 to 120.77]
Statistical Analysis 3: Comparison: Crizotinib CIC Fasted vs Crizotinib CIC Fed; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; Ratio of Adjusted means = 74.87, 90% CI 2-sided [67.55 to 82.98]

9. Secondary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUC [0 - ∞]) for Crizotinib Metabolite (PF-06260182)
Description: as for outcome 1
Time Frame: 0 (pre-dose), 1, 2, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96 and 144 hrs post crizotinib dose
Population: PK parameter analysis population included all randomized and treated participants who had at least 1 of the PK parameters of primary interest in at least 1 treatment period. Here, the 'N = 35' is signifying those participants who were evaluable for this measure at the specified time point for crizotinib CIC fed arm group.
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Crizotinib IRT Fasted | Crizotinib PIC Fasted | Crizotinib CIC Fasted | Crizotinib CIC Fed
Number analyzed (Participants) | 35 | 35 | 35 | 35
ng*hr/mL | 442.00 (221.96) | 402.10 (257.39) | 447.10 (248.23) | 341.80 (194.91)
Statistical Analysis 1: Comparison: Crizotinib IRT Fasted vs Crizotinib CIC Fasted; Natural log transformed AUC (0-∞) of PF-06260182 was analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. The adjusted mean differences and 90% CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios; Test type: Superiority or Other; Ratio of Adjusted means = 100.08, 90% CI 2-sided [90.46 to 110.73]
Statistical Analysis 2: Comparison: Crizotinib PIC Fasted vs Crizotinib CIC Fasted; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; Ratio of Adjusted means = 108.47, 90% CI 2-sided [98.03 to 120.02]
Statistical Analysis 3: Comparison: Crizotinib CIC Fasted vs Crizotinib CIC Fed; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; Ratio of Adjusted means = 76.59, 90% CI 2-sided [69.23 to 84.74]

10. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) for Crizotinib Metabolite (PF-06260182)
Time Frame: 0 (pre-dose), 1, 2, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96 and 144 hrs post crizotinib dose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Crizotinib IRT Fasted | Crizotinib PIC Fasted | Crizotinib CIC Fasted | Crizotinib CIC Fed
Number analyzed (Participants) | 35 | 35 | 35 | 36
ng/mL | 32.20 (12.48) | 29.74 (15.19) | 33.04 (12.12) | 23.64 (10.85)
Statistical Analysis 1: Comparison: Crizotinib IRT Fasted vs Crizotinib CIC Fasted; Natural log transformed Cmax of PF-06260182 was analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. The adjusted mean differences and 90% CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios; Test type: Superiority or Other; Ratio of Adjusted means = 102.11, 90% CI 2-sided [92.84 to 112.31]
Statistical Analysis 2: Comparison: Crizotinib PIC Fasted vs Crizotinib CIC Fasted; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; Ratio of Adjusted means = 108.87, 90% CI 2-sided [98.98 to 119.75]
Statistical Analysis 3: Comparison: Crizotinib CIC Fasted vs Crizotinib CIC Fed; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; Ratio of Adjusted means = 71.94, 90% CI 2-sided [65.46 to 79.05]

11. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) for Crizotinib Metabolite (PF-06260182)
Time Frame: 0 (pre-dose), 1, 2, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96 and 144 hrs post crizotinib dose
Population: as for outcome 2
Measure: Median (Full Range); unit: hr
Arm/Group | Crizotinib IRT Fasted | Crizotinib PIC Fasted | Crizotinib CIC Fasted | Crizotinib CIC Fed
Number analyzed (Participants) | 35 | 35 | 35 | 36
hr | 6.00 [4.00 to 8.02] | 6.00 [4.00 to 8.00] | 5.00 [4.00 to 10.00] | 6.00 [2.00 to 10.00]

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Crizotinib IRT Fasted | Crizotinib PIC Fasted | Crizotinib CIC Fasted | Crizotinib CIC Fed
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36 | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 21/36 | 24/36 | 20/36 | 21/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Crizotinib IRT Fasted (N=36) | Crizotinib PIC Fasted (N=36) | Crizotinib CIC Fasted (N=36) | Crizotinib CIC Fed (N=36)
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 9 | 13 | 13 | 13
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Epigastric discomfort (Gastrointestinal disorders) | 2 | 1 | 2 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 1 | 0 | 1 | 2
Gingivitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 5 | 10 | 2 | 5
Salivary hypersecretion (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Fatigue (General disorders) | 3 | 5 | 2 | 1
Feeling cold (General disorders) | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 3 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Joint sprain (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0
Dizziness postural (Nervous system disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 4 | 5 | 4 | 3
Paraesthesia (Nervous system disorders) | 1 | 1 | 1 | 1
Somnolence (Nervous system disorders) | 1 | 1 | 1 | 3
Hot flush (Vascular disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes